CLINICAL TRIAL: NCT01074034
Title: Clinical Research Evaluation of the ASSURE Device Atrial and Ventricular Tachyarrhythmia Therapies Registry
Brief Title: REASSURE AV Registry
Acronym: REASSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G040067
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Sudden Cardiac Death; Bradycardia
MeSH Terms: conditions — Death, Sudden, Cardiac; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AV Therapy Assessment group (Experimental): appropriate system performance of the atrial and ventricular tachyarrhythmia therapies in the ASSURE device
  Interventions: Device: AV Therapy Assessment-B301 investigational device

INTERVENTIONS:
Device: AV Therapy Assessment-B301 investigational device — Atrial and ventricular tachyarrhythmia therapy delivered by the B301 investigational device

SUMMARY:
Long term follow-up to monitor safety for patients implanted with a B301 ASSURE device.

DETAILED DESCRIPTION:
The Guidant ASSURE device is a fully featured pacemaker with additional atrial and ventricular tachyarrhythmia therapy features. The REASSURE AV study is a clinical evaluation to support approval of these features. This clinical study is intended to provide adequate performance data on two atrial tachyarrhythmia management features, namely the ATS and atrial ATP. In addition data will be collected to verify that the ventricular tachyarrhythmia rescue shock feature performs as intended in the clinical setting in combination with other pacemaker functions.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and capable of providing informed consent at an approved clinical investigational center, and able to attend the investigational center as required by the protocol
* Patient is implanted with an investigational B301 device as part of the REASSURE AV study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2006-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Alaska Heart Institute, Anchorage, Alaska
  - Northern California Heart Care, Larkspur, California
  - Orlando Regional Hospital, Orlando, Florida
  - Heart and Vascular Institute, St. Petersburg, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - St. Joseph Hospital, Savannah, Georgia
  - Good Samaritan Hospital, Downers Grove, Illinois
  - Heart Care Research Foundation, Merrionette Park, Illinois
  - St. Mary Medical Center, Hobart, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Louisville Cardiology Medical Group, Louisville, Kentucky
  - Medical Center Cardiologist Research, Louisville, Kentucky
  - Owensboro Mercy Health System, Owensboro, Kentucky
  - Ochsner Foundation Hospital, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Mary's Duluth Clinic, Duluth, Minnesota
  - St. Anthony's Medical Center, St Louis, Missouri
  - Sunrise Hospital & Medical Center, Las Vegas, Nevada
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Christ Hospital - Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Center For Cardiac Arrhythmias, Houston, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Chippenham Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B301 Device: B301 ASSURE Device: Atrial and ventricular tachyarrhythmia therapy delivered by the B301 investigational device
Period: Overall Study
Arm/Group | B301 Device
Started | 211
Completed | 205
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- AV Therapy Assessment Group: AV Therapy Assessment group, Atrial ATP and Atrial Therapy Suite (ATS)
  AV Therapy Assessment-B301 investigational device: Atrial and ventricular tachyarrhythmia therapy delivered by the B301 investigational device
  Ventricular tachyarrhythmia rescue shock feature
  AV Therapy Assessment-B301 investigational device: Atrial and ventricular tachyarrhythmia therapy delivered by the B301 investigational device
Arm/Group | AV Therapy Assessment Group
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 124
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 211

OUTCOME MEASURES:

1. Primary Outcome: Inappropriate Shock Free Rate
Description: Incidences of ventricular shock therapy up to three months post implant. Rescue shocks are intended for the treatment of cardiac arrhythmias detected in the ventricle at rates greater than 220 bpm, including arrhythmias that originate in the atria if they are conducted at rates greater than 220 bpm as this can be life threatening if persistent. Shocks delivered for other reasons will be considered inappropriate shocks.
Time Frame: Three months post-implant
Measure: Number; unit: % of shock free rates
Arm/Group | AV Therapy Assessment Group
Number analyzed (Participants) | 211
% of shock free rates | 97.2

2. Secondary Outcome: Conversion Success Rate up to Three Months Post-implant
Description: For a pacemaker patient who experiences a spontaneous high rate ventricular arrhythmia, the ASSURE device may provide rescue shocks, a faster and more effective response than external methods of rescue. Successful conversion of an episode is defined by conversion to either; sinus rhythm, sinus tachycardia or atrial pacing by one minute post therapy delivery.
Time Frame: Three months post-implant
Measure: Number; unit: % of conversion rates
Arm/Group | B301 Device
Number analyzed (Participants) | 22
% of conversion rates | 90.9

ADVERSE EVENTS:
Time Frame: Adverse events were collected from ICF signature until the last follow-up visit (three month follow up visit).
Description: An adverse event is defined as any undesirable clinical occurrence. This can be a subject health related complaint, change in health status, or product issue. A clinical event will not be reported if it existed at enrollment and continued unchanged thereafter unless the event worsened considerably and required additional medical or pharmacological treatment.
Arm/Group | B301 Device
All-Cause Mortality (participants affected / at risk) | 4/211
Serious Adverse Events (participants affected / at risk) | 52/211
Other Adverse Events (participants affected / at risk) | 17/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B301 Device (N=211)
Adverse reaction - General (General disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Aortic stenosis (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 5 (6)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Dislodgment - Elevated threshold - RV (Cardiac disorders) | 1 (1)
Dislodgment - Unable to capture - RA (Cardiac disorders) | 2 (2)
Dyspnea - Heart failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Early ERI - Random component failure (Cardiac disorders) | 1 (1)
Endocrine (Endocrine disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Extracardiac stimulation - RV (Cardiac disorders) | 1 (1)
Genitourinary (Reproductive system and breast disorders) | 5 (5) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Guidewire removal- femoral vein (Skin and subcutaneous tissue disorders) | 1 (1)
Head, eyes, ears, nose, throat (HEENT) (Eye disorders) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Hematological (Blood and lymphatic system disorders) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Hematoma - Pocket (<=30 days post-implant) (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
Inappropriate tachy therapy - SVT (Cardiac disorders) | 1 (1)
Integumentary (Skin and subcutaneous tissue disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Intermittent claudication (Cardiac disorders) | 1 (1)
Latching (General disorders) | 2 (2)
Migration (General disorders) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 7 (7) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Multiple symptoms (General disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Multi-system failure - Heart failure (Cardiac disorders) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral edema - Heart failure (Cardiac disorders) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Pulmonary edema - Heart failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Renal insufficiency - Heart failure (Renal and urinary disorders) | 1 (1)
Seroma - Pocket (<=30 days post-implant) (Blood and lymphatic system disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B301 Device (N=211)
Atrial fibrillation (Cardiac disorders) | 17 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other